CLINICAL TRIAL: NCT05843812
Title: "Evaluation of the Clinical Response to Magnesium Sulfate as an Adjuvant in Anesthesia in Bariatric Surgery"
Brief Title: Magnesium Sulfate in Bariatric Surgery
Acronym: MgSObs
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Lilia Edith Luque Esparza, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: C.B/01-04-23
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Anesthesia and Analgesia; Magnesium Sulfate; Bariatric Surgery Candidate
Keywords: Analgesia; Anesthesia; Magnesium Sulfate; Bariatric Surgery; Pain Postoperative; Receptors, N-Methyl-D-Aspartate
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood dna
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Magnesium sulphate: Patients who received preoperative infusion with magnesium sulfate as part of their anesthetic management
  Interventions: Drug: Magnesium Sulfate 10 MG/ML
- No Magnesium sulphate: Patients who did not receive preoperative magnesium sulfate infusion as part of their anesthetic management

INTERVENTIONS:
Drug: Magnesium Sulfate 10 MG/ML — Patients who received preoperative infusion with magnesium sulfate as part of their anesthetic management
  Groups: Magnesium sulphate

SUMMARY:
Weight loss surgery, also known as bariatric surgery, has been around since the 1950s and since its inception has been shown to successfully achieve significant and sustainable weight loss in a large number of patients who undergo this intervention, as well , if a beneficial impact is observed in the management of metabolic disorders, such as type 2 diabetes mellitus and hyperlipidemia.

After bariatric surgery, patients are at risk of narcotic-related side effects.(2) Because of this, pain management strategies must be implemented to reduce the consumption of narcotic medications. Some studies have reported that a multimodal analgesic regimen can reduce the consumption of postoperative narcotics, as well as the therapy requirements to control postoperative nausea and vomiting.

It has also been reported that excess body mass is associated with changes in mineral levels in the body, particularly hypomagnesemia , a condition that is also common in hospitalized patients (Hansen & Bruserud 2018), and has a high incidence in the perioperative environment.

Magnesium sulfate (MgSO4) has multiple desirable effects in an anesthetic procedure. It is an antagonist of the N-methyl-d-aspartic acid (NMDA) receptor, which is why it produces an analgesic effect related to the prevention of central sensitization caused by peripheral tissue injury. In addition, other relevant clinical effects of MgSO4 have been reported in anesthesiology, such as its effect as a CNS depressant, modulation of the hemodynamic response, reduction of the intraoperative requirements of anesthetics, analgesics, and muscle relaxants. As well as the potentiation of the effect of non-depolarizing muscle relaxants.

The role of magnesium in the body and its pharmacological properties continue to be studied and knowledge of its pharmacological, clinical and physiological characteristics has become essential for the anesthesiologist.

There are no previous studies that allow establishing an optimal therapeutic scheme considering all the perioperative clinical effects of MgSO4 and that evaluate the role of genetic variability in pain perception and response to treatment in bariatric surgery.

DETAILED DESCRIPTION:
A total of 104 participants, men and women over the age of 18, scheduled for bariatric surgery, will be included. After accepting and signing the informed consent, a brief preoperative clinical history will be taken, a peripheral blood sample will be taken to determine preoperative serum Ca2+ and Mg2+, and to analyze polymorphic variants related to pain perception and the pharmacokinetics of analgesics. The clinical effect of MgSO4 on analgesia (EVAD), hemodynamic stability (BP and HR), intubation conditions, and satisfaction with anesthetic recovery will be evaluated. The presence of adverse reactions to anesthesia (nausea, vomiting, chills, pruritus, urinary retention, arrhythmias, laryngeal or bronchial spasm) and total doses of drugs used during the perioperative period will be recorded. All patients will undergo a standard pre, trans and postoperative protocol and according to the treatment received with MgSO4 as part of their anesthetic management or not, they will be assigned to the corresponding group (MgSO4/ No MgSO4). All the data will be collected in an Excel database, for subsequent analysis in SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for bariatric surgery under general o anesthesia at Hospital universitario de la Facultad de Medicina de la Universidad Autonoma de Coahuila
* Physical state ASA 2 y 3
* Acceptance and signing of the informed consent.

Exclusion Criteria:

* Treatment with calcium or magnesium channel blockers
* Drug use or alcoholism referred by the patient in the questioning
* Neurological diseases
* Myopathy
* Intracardiac block
* Renal insufficiency
* Liver failure
* Pregnancy
* Hematological disorders
* Contraindications to the use of magnesium sulfate (hypersensitivity to the active principle or to any of the excipients, concomitant use with quinidine derivatives, tachycardia, heart failure, myocardial injury, infarction).

Elimination criteria:

* Survey with incomplete data corresponding to the study variables.
* Revocation of informed consent or decision to withdraw by of the patient.
* Loss to follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Men and women over the age of 18, scheduled for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in postoperative analgesia over 24 hours | [Time Frame: 15 minutes after coming out of anesthesia, 2, 4, 6 and 24 hours after coming out of anesthesia]
  Postoperative pain intensity reported by the participant using the visual analog scale after bariatric surgery
Time to first request for pain reliever | [Time Frame: 24 hours after departure from anesthesia]
  Time (minutes) to request analgesia after coming out of bariatric surgery
Hemodynamic stability | [Time Frame: 180 minutes intraoperatively]
  Changes in heart rate (beats per minute) and mean systemic arterial pressure (mmHg) intraoperatively after or during bariatric surgery were combined to report hemodynamic stability.
  Measurements of heart rate and mean arterial pressure will be added to arrive at a reported value (hemodynamic stability: yes or no).
  Changes in heart rate (beats per minute) and mean systemic arterial pressure (mmHg) less than 20% with respect to baseline values will be considered as criteria for hemodynamic stability, without the need to administer atropine, ephedrine or other positive chronotropic agents and / or vasoactive agents.
Interaction with neuromuscular blockers (BNM): Onset time | [Time Frame: 180 minutes intraoperatively]
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Onset time (OT): Time elapsed from the administration of BNM to obtaining a depression in the monitored motor response of between 80 to 100% with the T1 stimulus pattern of TOF.
Interaction with neuromuscular blockers (BNM):Clinical effect time | [Time Frame: 180 minutes intraoperatively]
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Clinical effect time: Time elapsed from administration of BNM until 25% is recovered in the monitored motor response measured with TOF as T1> 25% or ST> 25%.
Interaction with neuromuscular blockers (BNM): Recovery index (RI) | [Time Frame: 180 minutes intraoperatively]
  Parameters measured per train of four after administration of the non-depolarizing muscle relaxant according to the parameters established in the current guidelines for good clinical research practices in pharmacodynamic studies of neuromuscular blocking agents II:
  - Recovery index (RI): Time elapsed between recovery of 25% and 75% of T1 from TOF.

SECONDARY OUTCOMES:
Adverse reactions to magnesium sulfate | [Time Frame: From the start of the magnesium sulfate infusion until 24 hours after leaving anesthesia]
  Adverse reactions to the perioperative administration of parenteral magnesium sulfate that derive from magnesium poisoning or alterations in the administration site.
  Administration site alterations (injection site pain, hypothermia, vasodilation with a sensation of heat).
  Nervous system (loss of tendon reflex, headache, dizziness, coma, drowsiness and confusion, CNS depression, respiratory paralysis).
  Cardiovascular system (circulatory collapse, arrhythmias, cardiac arrest).
  Respiratory system (respiratory depression secondary to neuromuscular block).
  Gastrointestinal system (nausea and vomiting).
  Musculoskeletal and connective tissue system (muscle weakness).
  Others (problems with speech, vision, excessive sweating, thirst, or others not reported).
Adverse reactions to anesthesia | [Time Frame: 180 minutes intraoperatively up to 24 hours after discharge from anesthesia]
  Side and adverse effects associated with the use of anesthetic drugs.
  Nausea, vomiting, itching, chills, urinary retention, arrhythmias, laryngeal or bronchial spasm.
Number of participants carrying polymorphisms related to perioperative clinical response to magnesium sulfate | [Time Frame: During the 2-year duration of the study]
  Determination of polymorphisms related to the pharmacokinetics of opioids (gene CYP3A4/*16, CYP3A4/*1B), the NMDA receptor (GENE NR1/GRIN1, NR2/GRIN2A, NR2B/GRIN2B, NR3A/GRIN3A, NR3B/GRIN3B), and magnesium transporters (gene CNNM2, TRPM6, SLC41A1, SLC41A2).
Conditions for endotracheal intubation | 5 minutes after the administration of BNM
  Evaluation of the conditions for orotracheal intubation. Use a qualitative scoring system. The factors that are taken into consideration are: ease of laryngoscopy, position and / or movement of the vocal cords and reaction to intubation.
Consumption of intraoperative analgesics | 180 minutes intraoperatively
  Consumption of analgesics (μg of fentanyl) intraoperatively in induction and / or maintenance in each group of patients.
Postoperative analgesic consumption | From exit from anesthesia up to 24 hours
  Consumption of opioid analgesics (evaluated as mg morphine equivalents) postoperatively
Consumption of neuromuscular relaxant | 180 minutes intraoperatively
  Consumption of neuromuscular relaxant (mg of cisatracurium) intraoperatively in intubation and / or maintenance after / during bariatric surgery, in each study group.
Hypnotic use | 180 minutes intraoperatively
  Hypnotic consumption (mg of propofol) intraoperatively in intubation and / or maintenance after / during bariatric surgery, in each study group.
Satisfaction in recovery from anesthesia | 24 hours after departure from anesthesia
  The overall satisfaction of the patients was evaluated the day after surgery using the IOWA scale (Dissatisfied: -3-2-1, Satisfied + 1 + 2 + 3) after bariatric surgery.

OTHER OUTCOMES:
Serum magnesium | Before IV infusion of MgS04 and 24 hours after coming out of anesthesia
  Serum magnesium concentrations(mg / dL)
Intracellular magnesium | Before IV infusion of MgS04 and 24 hours after coming out of anesthesia
  Magnesium content in erythrocyte cells

CONTACTS AND LOCATIONS:
Locations (1):
- Lilia Edith Luque-Esparza, Gómez Palacio, Durango, Mexico

IPD SHARING:
Plan to Share IPD: Undecided